CLINICAL TRIAL: NCT06435702
Title: A Prospective Observational Cohort Study of Efficacy and Safety of Darolutamide in Combination With Androgen-Deprivation Therapy in Prostate Cancer Patients With Lymph Node-positive After Radical Prostatectomy
Brief Title: Efficacy and Safety of Darolutamide in Combination With Androgen-Deprivation Therapy in Prostate Cancer Patients With Lymph Node-positive After Radical Prostatectomy: A Prospective Observational Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: LM2023526
Record Dates: First submitted 2024-05-26; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: Lymph Node-positive; Prostate Cancer; Radical Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — darolutamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Darolutamide in addition to androgen deprivation therapy: Darolutamide 600mg twice daily. The ADT regimen was either a gonadotropin-releasing hormone analog agonist or a gonadotropin-releasing hormone antagonist.The ADT administration type, frequency, and dose were determined by the investigator.
  Interventions: Drug: Darolutamide in addition to androgen deprivation therapy
- androgen deprivation therapy only: The ADT regimen was either a gonadotropin-releasing hormone analog agonist or a gonadotropin-releasing hormone antagonist.The ADT administration type, frequency, and dose were determined by the investigator.
  Interventions: Drug: androgen deprivation therapy only

INTERVENTIONS:
Drug: Darolutamide in addition to androgen deprivation therapy — Darolutamide 600mg twice daily. The ADT regimen was either a gonadotropin-releasing hormone analog agonist or a gonadotropin-releasing hormone antagonist.The ADT administration
  Groups: Darolutamide in addition to androgen deprivation therapy
Drug: androgen deprivation therapy only — The ADT regimen was either a gonadotropin-releasing hormone analog agonist or a gonadotropin-releasing hormone antagonist.The ADT administration type, frequency, and dose were determined by the investigator.
  Groups: androgen deprivation therapy only

SUMMARY:
This study is an open, prospective, single-center observational clinical study to evaluate the efficacy and safety of immediate adjuvant ADT with darotarolimide in the treatment of patients with positive lymph nodes after radical prostatectomy for prostate cancer.

DETAILED DESCRIPTION:
This study is an open, prospective, single-center observational clinical study to evaluate the efficacy and safety of immediate adjuvant ADT with darotarolimide in the treatment of patients with positive lymph nodes after radical prostatectomy for prostate cancer. The study evaluates the efficacy of immediate adjuvant ADT with darotarolimide in patients with positive lymph nodes after radical prostatectomy for prostate cancer, using time to achieve CRPC as the primary study endpoint. OS will be examined in all patients after the primary study endpoint is achieved and will serve as the key secondary study endpoint. It is planned to enroll 108 patients with positive lymph nodes after radical prostatectomy for prostate cancer. It is divided into a screening period, a treatment period and a follow-up period. Patients will enter the screening period from the time they sign the informed consent form, and those who have been evaluated and qualified in the screening period will be entered into the study. Patients eligible for enrollment will receive 2 years of ADT treatment or ADT treatment + darotarotide adjuvant therapy with or without combination radiotherapy at the investigator's discretion.

ELIGIBILITY:
Inclusion Criteria:

* 1. patients voluntarily enrolled in the study and signed an informed consent form; 2. aged 18-80 years (including 18 and 80 years), male; 3. diagnosed with prostate adenocarcinoma by pathology or cytology; 4. Eastern Cooperative Oncology Group (ECOG) Physical Status (PS) score 0-1. 5. patients who have undergone radical prostatectomy (RP) and pelvic lymph node dissection (PLND) without non-regional lymph node metastasis, bone metastasis, or metastasis to other sites (e.g., visceral metastasis) as confirmed by conventional imaging (bone imaging, CT, or MRI) or PSMA PET/CT 6. have positive postoperative pathologic lymph nodes (pN1); 7. with their consent and have signed an informed consent form.

Exclusion Criteria:

* Patients will not be enrolled if they have any of the following:

  1. have histologic features of neuroendocrine differentiation or small cell carcinoma;
  2. have received prior treatment for prostate cancer: postoperative systemic therapy including ADT for >3 months, conventional endocrine therapy (e.g., flutamide, bicalutamide) for >3 months, novel endocrine therapy (e.g., dalotamide, abiraterone, abatacept, enzalutamide), chemotherapy (e.g., docetaxel), immunotherapy, and targeted therapies
  3. Inability to tolerate Darotamine or ADT treatment;
  4. persons who are allergic or have a known history of allergy to darotarolimide or ADT;
  5. other conditions that the investigator considers inappropriate for inclusion.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients with non-metastatic prostate cancer who underwent radical prostatectomy with positive pathologic lymph nodes
Sampling Method: Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to CRPC | Time from initiation to the occurrence of PSA progression or imaging progression, whichever occurs first.
  castrate resistant prostate cancer

SECONDARY OUTCOMES:
MFS | Time to metastasis or death confirmed from enrollment imaging, whichever occurred first
  metastasis-free survival
rPFS | Time from initiation to imaging progression or death from any cause, whichever occurs first
  radiography Progression-Free-Survival
PSA-PFS | Time from initiation to PSA progression or death, whichever occurs first
  radiography Progression-Free-Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China